CLINICAL TRIAL: NCT04244955
Title: Observational Study Evaluating the Psychic Impact of the Diagnostic Announcement and Care for Children Treated for Cancer
Acronym: IPSYLON
Status: Terminated | Type: Observational
Why Stopped: Investigator's decision
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET19-292 IPSYLON
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Semi-directive interviews — The interviews, carried out by the child psychiatrist, will be semi-directive and short (15 to 30 minutes) one-on-one with the child or adolescent so that the presence of the parents does not influence the responses. The CPTS-RI index, which has 20 questions, will be filled, as well as other questions to understand what is problematic for the child.

SUMMARY:
The cancer diagnostic announcement and cancer care are both physical and psychological highlights. The main objective is to analyze significant psychological difficulties in children aged 6 to 16 treated for cancer.

DETAILED DESCRIPTION:
Symptoms of post traumatic stress disorder in young children are often underdiagnosed because the criteria of DSM-IV and ICD-10 are not suitable for these children. These symptoms are nightmares, sleep problems, compulsive and joyless gambling, regression, hyper attention, anxiety over new separation, and new fears. It is also known that the disorders are readily more marked at the start of treatment and then subside throughout the first year. Some may appear afterwards after treatment.

To our knowledge, no study has evaluated the prevalence of mental disorders linked to diagnosis and care during treatment and their link with the practice of care. This study will focus on disorders during treatment. We will study the psychic impact of the announcement of diagnosis and care, whether they belong to the traumatic dimension or not. For this, we will use the validated French version of the Child Post-Traumatic Stress Reaction Index (CPTS-RI) scale. It is the most widely used scale in clinical research of trauma and reactive mental disorders in children 6 to 16 years of age. We will also assess the most disturbing elements for the child and the main clinical manifestations found in order to improve the detection of mental disorders and the care support for these children.

This research will allow us to assess the prevalence of mental disorders in connection with the care practiced within the Institute of Pediatric Hematology and Oncology (IHOPe) and, subsequently, to establish a another intervention research protocol to improve our practices and the care of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 6 to 16 years;
* Patient diagnosed for a malignant pathology for at least one month and maximum 2 months;
* Patient treated at the IHOPe;
* Non-opposition of the parents and the child under study.

Exclusion Criteria:

* Difficulty speaking and understanding French;
* Patient who is not able to express himself because the somatic medical conditions do not allow a verbal exchange.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric cancer
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Analyze of significant psychological difficulties in children aged 6 to 16 | 30 minutes
  Score at the Child Post-Traumatic Stress Reaction Index (CPTS-RI) questionnaire. A score strictly greater than 24 on the CPTS-RI questionnaire will be considered clinically significant for the primary endpoint

SECONDARY OUTCOMES:
Evaluation of the most disturbing elements for the child and the main clinical manifestations found. | 30 minutes
  Most disturbing elements for the child (since the start of care and in invasive and / or repeated care) and the main clinical manifestations found during the semi-directive interviews, carried out by the child psychiatrist.
Collection of the opinion of the caregivers (doctors, nurses) of each patient on the psychic impact of care on the child. | 30 minutes
  Rating of the level of difficulty similar to the CPTS-RI scale: none, mild, moderate, severe or very severe.
Evaluation of the agreement between the levels of difficulty rated by the child and his caregivers. | 30 minutes
  Measure of agreement between the two evaluations using Kappa coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Elodie SAVOURÉ, M.D, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No